CLINICAL TRIAL: NCT03664518
Title: A Multicenter Single-arm Study to Evaluate the Efficacy and Safety of Eltrombopag for Immune Thrombocytopenia in Chinese Patients With Chronic HBV Infection
Brief Title: to Evaluate the Efficacy and Safety of Eltrombopag for Immune Thrombocytopenia With Chronic HBV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Novartis (Industry); Qilu Hospital of Shandong University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Tianjin First Central Hospital (Other); Tianjin Medical University Second Hospital (Other); Henan Cancer Hospital (Other Government); The Second Hospital of Hebei Medical University (Other); North China University of Science and Technology (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018006
Record Dates: First submitted 2018-08-26; First posted 2018-09-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2023-08

CONDITIONS: Thrombocytopenia Purpura; Chronic HBV Infection
MeSH Terms: conditions — Purpura, Thrombocytopenic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eltrombopag (Experimental): 58 enrolled patients are picked up to take eltrombopag at the indicated dose.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — subjects will initiate treatment with 25 mg eltrombopag. Platelet counts is obtained weekly and dose adjustment should be done according to platelet counts. and maximum dose should not exceed 75 mg daily. Subjects whose platelet count between 50~150×109/L，the eltrombopag dose Maintain. platelet count between 150~250×109/L, need to reduce the dose of eltrombopag to the next lower dose or lower frequency. Subjects whose platelet count exceeds 250×109/L at any point during the treatment period, must have eltrombopag interrupted and increase the frequency of platelet monitoring to twice weekly, until platelet counts fall below 100×109/L.

SUMMARY:
Primary Objective: To evaluate the efficacy of 6-week Eltrombopag to treat immune thrombocytopenia with chronic hepatitis B virus infection. Secondary Objective: To evaluate the efficacy and safety of 6-week and 22-week Eltrombopag to treat immune thrombocytopenia with chronic hepatitis B virus infection.

DETAILED DESCRIPTION:
This is a single-arm phase II study to evaluate the efficacy and safety of Eltrombopag to treat immune thrombocytopenia with chronic hepatitis B virus infection.

This study includes two stages. In Stage 1 (Week 1 to Week 6), the short-term efficacy, safety and tolerability of Eltrombopag is evaluated. At the end of Stage 1, the subjects who can benefit from Eltrombopag treatment (platelet count ≥30×109/L at least once and a 2-fold increase from baseline platelet count without rescue therapy, with no bleeding) can enter a 16-week prolonged stage (Stage 2) to evaluate longer-term efficacy and safety.

The starting dose of Eltrombopag is 25 mg once daily, and the dose may be increased by 25 mg once daily according to protocol if the desired platelet response (>50×109/L) is not achieved. The daily dose should not exceed 75 mg.

In Stage 1, weekly visits are required during the first 6 weeks of the study. In Stage 2, platelet counts will be obtained weekly during dose adjustment and every 4 weeks following establishment of a stable dose of Eltrombopag (stable dose is defined as the dose which remains unchanged for at least 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Subject is ≥18 years old.
* Diagnosis of HBV-infection duration for at least 6 months prior to the study and have a platelet count of <30 ×109/L on Day 1 (or within 48 hours prior to dosing on Day 1).
* Complete blood count results: white blood cells, absolute neutrophils count and hemoglobin are within the laboratory normal range, but abnormalities caused by HBV infection can be accepted.
* Subject is practicing an acceptable method of contraception. Women of childbearing potential must have a negative serum pregnancy test in the whole study.

Exclusion Criteria:

* Liver cirrhosis (LC) defined as any of the following:

  1. Any symptom or sign typical of hepatic decompensation: including but not limited to ascites, splenomegaly, dilation of periumbilical collateral veins, hepatic encephalopathy
  2. Child-Pugh class B to C Biopsies are not required either for confirmation or for exclusion of LC, considering the high bleeding risk in these patients.
* Positive serology for HIV, hepatitis C virus (HCV), and/or hepatitis D virus (HDV).
* Pregnancy or lactation period.
* History of alcohol/drug abuse or dependence within 12 months of the study.
* History of thrombosis.
* The serum chemistry results exceed the upper laboratory normal range by more than 20%; except AST, ALT, GGT, ALP of CTCAE grade 1.
* Bone marrow examination conducted within 4 weeks prior to first dose reported an abnormal result, which in the opinion of the investigator makes the subject unsuitable for participation in the study.
* Pre-existing cardiac disease, including congestive heart failure of New York Heart Association [NYHA] Grade III/IV, arrhythmia requiring treatment or myocardial infarction within the last 6 months. No arrhythmia known to increase the risk of thrombotic events (e.g. atrial fibrillation), or patients with a QT >450msec or QTc > 480 for patients with a Bundle Branch Block.
* Subject has consumed aspirin, aspirin-containing compounds, salicylates, anticoagulants, quinine or non-steroidal anti-inflammatories (NSAIDs) for >3 consecutive days within 2 weeks prior to the study start and until the end of the study.
* Non-compliant patient
* Reluctance to take effective contraceptive measures during the trial
* History of solid organ or bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a platelet count ≥ 50×109/L at Day 43 | 6 weeks
  The proportion of subjects with a platelet count ≥ 50×109/L at Day 43 after the first 6 weeks of Eltrombopag treatment (Stage 1)

SECONDARY OUTCOMES:
Response rate of treatment | 22 weeks
  Response rate including: a) the proportion of subjects achieving platelet counts ≥ 50×109/L at least once during the first 6 weeks (stage 1); b) the proportion of subjects whose platelet counts ≥ 30×109/L and at least two times of baseline platelet count at least once during the treatment.
Bleeding in two stages | 22 weeks
  according to the WHO bleeding grades to estimate the incidence and severity of bleeding symptoms during the treatment.
The duration time with Platelet count ≥ 50×109/L | 22 weeks
  Total duration of time a subject had a platelet count ≥ 50×109/L during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: lei zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Ethics Committee of Blood disease hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.

REFERENCES:
- [Background] Ott JJ, Stevens GA, Groeger J, Wiersma ST. Global epidemiology of hepatitis B virus infection: new estimates of age-specific HBsAg seroprevalence and endemicity. Vaccine. 2012 Mar 9;30(12):2212-9. doi: 10.1016/j.vaccine.2011.12.116. Epub 2012 Jan 24. PMID 22273662
- [Background] Zhang Y, Zhang H, Elizabeth A, Liu XQ. Epidemiology of hepatitis B and associated liver diseases in china. Chin Med Sci J. 2013 Jan;27(4):243-8. doi: 10.1016/s1001-9294(13)60009-7. PMID 23294591
- [Background] Toghill PJ, Green S, Ferguson F. Platelet dynamics in chronic liver disease with special reference to the role of the spleen. J Clin Pathol. 1977 Apr;30(4):367-71. doi: 10.1136/jcp.30.4.367. PMID 853132
- [Background] Aref S, Mabed M, Selim T, Goda T, Khafagy N. Thrombopoietin (TPO) levels in hepatic patients with thrombocytopenia. Hematology. 2004 Oct-Dec;9(5-6):351-6. doi: 10.1080/10245330400010620. PMID 15763973
- [Background] Afdhal N, McHutchison J, Brown R, Jacobson I, Manns M, Poordad F, Weksler B, Esteban R. Thrombocytopenia associated with chronic liver disease. J Hepatol. 2008 Jun;48(6):1000-7. doi: 10.1016/j.jhep.2008.03.009. Epub 2008 Mar 31. PMID 18433919
- [Background] Bussel JB, Marks KM. How effective is eltrombopag for the treatment of thrombocytopenia in patients with HCV infection? Nat Clin Pract Gastroenterol Hepatol. 2008 Aug;5(8):424-5. doi: 10.1038/ncpgasthep1185. Epub 2008 Jul 8. No abstract available. PMID 18607406
- [Result] Yang R, Li J, Jin J, Huang M, Yu Z, Xu X, Zhang X, Hou M. Multicentre, randomised phase III study of the efficacy and safety of eltrombopag in Chinese patients with chronic immune thrombocytopenia. Br J Haematol. 2017 Jan;176(1):101-110. doi: 10.1111/bjh.14380. Epub 2016 Oct 13. PMID 27734464
- [Result] Bussel JB, Cheng G, Saleh MN, Psaila B, Kovaleva L, Meddeb B, Kloczko J, Hassani H, Mayer B, Stone NL, Arning M, Provan D, Jenkins JM. Eltrombopag for the treatment of chronic idiopathic thrombocytopenic purpura. N Engl J Med. 2007 Nov 29;357(22):2237-47. doi: 10.1056/NEJMoa073275. PMID 18046028
- [Result] Giannini EG, Afdhal NH. Eltrombopag in patients with chronic liver disease. Expert Opin Pharmacother. 2013 Apr;14(5):669-78. doi: 10.1517/14656566.2013.775249. Epub 2013 Mar 4. PMID 23452139